CLINICAL TRIAL: NCT01205737
Title: A Phase Ib, Double Blind RCT to Evaluate and Compare the PK, PD and Safety of MabThera® With TL011, in Combination With CHOP, in Subjects With CD20+ DLBCL
Brief Title: A Double-blind, Randomized Controlled Study in CD20-positive Diffuse B Cell Non-Hodgkin's Lymphoma Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NHL-TL011-102
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: DLBCL
Keywords: DLBCL; pharmacokinetics; pharmacodynamics
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TL011 (Experimental)
  Interventions: Biological: TL011
- MabThera® (Active Comparator)
  Interventions: Biological: Rituximab

INTERVENTIONS:
Biological: TL011 — 375 mg/m2 iv every 3 weeks for 8 cycles
  Arms: TL011
Biological: Rituximab — 375 mg/m2 iv every 3 weeks for 8 cycles
  Arms: MabThera®

SUMMARY:
This is a prospective international, multi-center, randomized, double-blind controlled study designed to assess and compare the pharmacokinetics, pharmacodynamics and the safety of MabThera® and TL011, in combination with CHOP in previously untreated patients with diffuse large B cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed subjects with a confirmed pathologic diagnosis of diffuse large B cell non-Hodgkin's lymphoma (DLBCL) based on the 2008 World Health Organization classification.

  2.CD20+ lymphoma cells at screening
* 18-80 (inclusive) years of age at screening
* Ann Arbor Stages I-IV at screening
* Any IPI score at screening
* ECOG good performance status (0-2) at screening
* Willing and able to provide written informed consent prior to performing study procedures
* Women of childbearing potential must use effective contraceptive methods starting from screening and until 12 months following the last infusion..

Exclusion Criteria:

1. Any lymphoma other than CD20+ DLBCL
2. History of indolent lymphoma
3. DLBCL with central nervous system or meningeal involvement
4. Primary gastrointestinal (MALT) lymphoma
5. Bulky disease>10 cm diagnosed by imaging at screening
6. Bone marrow involvement > 25% according to bone marrow biopsy at screening
7. Subjects previously treated with chemotherapy, radiotherapy, immunotherapy or experimental therapies for lymphoma or other malignancy
8. Hypersensitivity to active ingredients, excipients (sodium citrate, polysorbate 80, sodium chloride, sodium hydroxide, hydrochloric acid, water for injections) and murine proteins
9. Active uncontrolled infection (viral, bacterial or fungal infection) requiring systemic therapy at screening and/or at baseline visit.
10. A documented history of recurrent or chronic clinically significant infection (viral, bacterial or fungal infection)
11. Subjects with a history of tuberculosis or active tuberculosis at screening.
12. Immunodeficiency syndrome or Human immunodeficiency virus (HIV) seropositivity
13. Positive Hepatitis B surface antigen or antibodies to Hepatitis C
14. History of other cancer within the past 5 years except curatively treated non-melanoma skin cancer or in situ carcinoma of uterine cervix
15. Any major surgical procedure within 12 weeks prior to screening and between screening and baseline
16. Immunization with live viral vaccines less than 4 weeks prior to first study drug infusion, and/or planned live viral vaccination during study period.
17. Known allergic reactions against foreign proteins
18. Subjects for whom 8 cycles of CHOP might be problematic, and have the following findings/conditions, should not be enrolled:

    * Cardiac contra-indication to doxorubicin: Left ventricular ejection fraction (LVEF) < 50% according to multi-acquisition gated (MUGA) scan or 2D Echocardiogram at screening
    * Neurologic contra-indication to vincristine: (e.g., peripheral neuropathy)
    * Abnormal hepatic function at screening and/or baseline
    * AST/ALT ≥ 3 x upper normal value (ULN) or ≥ 5 x ULN in the presence of DLBCL involvement of the liver
    * Bilirubin ≥ 2 x ULN or ≥ 5 x ULN in the presence of DLBCL involvement of the liver
    * Abnormal renal function at screening and/or baseline
    * Serum creatinine ≥ 2 x ULN
    * Abnormal bone marrow function at screening and/or baseline
    * Platelets < 100x109/L
    * Neutrophils < 1.5x109/L
    * Hb < 9g/dL
19. Any other serious active disease or co-morbid medical condition (according to the investigator's decision and information provided in the Investigator Brochure of TL011)
20. Subjects who, according to the investigator, are likely to be non-compliant or uncooperative during the study.
21. Pregnant or lactating women or women that intend to get pregnant during study or within 12 months following the last infusion.
22. Treatment with any investigational drug within 90 days before planned first cycle of chemotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2010-09; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
AUC during a dosing interval for Rituximab | 21 weeks

SECONDARY OUTCOMES:
PK and PD parameters | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, PhD, Principal Investigator — Hospital Universitario Puerta de Hierro
Locations (41):
- Bulgaria (5):
  - Teva Investigational Site 59005, Pleven
  - Teva Investigational Site 59003, Plovdiv
  - Teva Investigational Site 59001, Sofia
  - Teva Investigational Site 59002, Sofia
  - Teva Investigational Site 59004, Varna
- Estonia (2):
  - Teva Investigational Site 55001, Tallinn
  - Teva Investigational Site 55002, Tartu
- Teva Investigational Site 35066, Paris, France
- Teva Investigational Site 51026, Debrecen, Hungary
- Italy (2):
  - Teva Investigational Site 30001, Florence
  - Teva Investigational Site 30002, Napoli
- Latvia (3):
  - Teva Investigational Site 56002, Daugavpils
  - Teva Investigational Site 56001, Riga
  - Teva Investigational Site 56003, Riga
- Teva Investigational Site 53010, Warsaw, Poland
- Russia (12):
  - Teva Investigational Site 50011, Arkhangelsk
  - Teva Investigational Site 50001, Chelyabinsk
  - Teva Investigational Site 50006, Kazan'
  - Teva Investigational Site 50014, Kursk
  - Teva Investigational Site 50005, Moscow
  - Teva Investigational Site 50009, Moscow
  - Teva Investigational Site 50010, Moscow
  - Teva Investigational Site 50003, Novosibirsk
  - Teva Investigational Site 50017, Pyatigorsk
  - Teva Investigational Site 50012, Saint Petersburg
  - Teva Investigational Site 50015, Tomsk
  - Teva Investigational Site 50004, Yekaterinburg
- Spain (6):
  - Teva Investigational Site 31005, Elche-Alicante
  - Teva Investigational Site 31006, Las Palmas de Gran Canaria
  - Teva Investigational Site 31002, Madrid
  - Teva Investigational Site 31001, Majadahonda-Madrid
  - Teva Investigational Site 31003, Valencia
  - Teva Investigational Site 31004, Valencia
- Ukraine (8):
  - Teva Investigational Site 58011, Cherkasy
  - Teva Investigational Site 58013, Dnipropetrovsk
  - Teva Investigational Site 58014, Donetsk
  - Teva Investigational Site 58017, Khmelnytskyi
  - Teva Investigational Site 58010, Kyiv
  - Teva Investigational Site 58012, Kyiv
  - Teva Investigational Site 58015, Kyiv
  - Teva Investigational Site 58016, Simferopol